CLINICAL TRIAL: NCT01160224
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Compare GW766944 (an Oral CCR3 Receptor Antagonist) Versus Placebo in Patients With Asthma and Sputum Eosinophilia.
Brief Title: Oral GW766944 (Oral CCR3 Antagonist)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 114312
Record Dates: First submitted 2010-06-10; First posted 2010-07-12 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Asthma
Keywords: Asthma; CCR3 receptor antagonists; GW766944
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GW766944 (Active Comparator): This is the active drug (GW766944)
  Interventions: Drug: GW766944
- Placebo (Placebo Comparator): Placebo Arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GW766944 — Drug: GW766944 (Active Drug Treatment)
  Arms: GW766944
Other: Placebo — This is placebo to match.
  Other Names: Placebo Treatment
  Arms: Placebo

SUMMARY:
GW766994 is a selective, competitive antagonist of the human CC chemokine receptor-3 (CCR3). It is proposed that the inhibition of the CCR3 receptor may provide a treatment for airway inflammation such as in asthma. This will be a double-blind, placebo controlled, parallel group study being conducted to evaluate the effects of GW766994 in subjects with mild-moderate asthma who have high sputum eosinophilia. The primary objective is to compare the effects of GW766994 to placebo on sputum eosinophils.

DETAILED DESCRIPTION:
This will be a multi-centre study. This is a randomized, double-blind, placebo-controlled, parallel-group study, in patients with asthma and eosinophilic bronchitis. Subjects with asthma will be atopic and not on oral prednisone. Inhaled corticosteroids are allowed if on stable dose. All subjects will receive a 5 day course of 30mg daily of oral prednisone after one week stopping study drug.

All subjects will attend screening (Visit 1) at which their eligibility for inclusion will be assessed. Eligible subjects will be randomized to receive either 300 mg of GW766994 twice daily or matching placebo at Day 1 (Visit 2) and will be stratified according to the subject's sputum eosinophil count at Visit 1. Treatment will be 10 days of oral dosing, and subjects will participate in a Day 7 or 8 visit (Visit 3), Day 10 visit (Visit 4 - End of Treatment), followed by a 1 week wash out period (Visit 5 -Follow Up Visit). At Visit 5, all subjects will be given 30 mg oral daily prednisone for 5 days and subjects to return to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22.

Pharmacodynamic assessments will include both sputum and blood biomarkers and spirometry.

Safety will be assessed by vital sign measurement, electrocardiogram, clinical laboratory tests (hematology, chemistry & urinalysis), clinical monitoring and adverse event reporting. Pharmacokinetic samples will be collected from each subject according to the sample schedule in the timing and events table.

Study will involved sputum biology (progenitors, cell counts). Study will be conducted in Canada only.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma (>12% improvement in FEV1 with a bronchodilator or PC20 methacholine less than 8 mg/ml) documented within the past 2 years.
* Males and females aged ≥18-75 years inclusive.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Child-bearing potential and agrees to use one of the contraception methods listed in Section 9.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 2 days after the last dose of GW766994.
* Non smoker. Current smokers with a with a pack history of less than 10 years may be enrolled into the study. Subjects who only use chewing tobacco products may be enrolled at the discretion of the Investigator and after consultation with the GSK medical monitor.
* Sputum eosinophils >4.9%.
* AST, ALT, alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QTcB or QTcF < 450 msec assessed within 6 months of the screening visit.
* To be eligible, female patients must have a negative urine pregnancy test.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The subject is able to understand and comply with protocol requirements, instructions and protocol- stated restrictions.

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination, or ECG.
* Current smokers.
* Subjects unable to produce a technically acceptable sputum sample.
* Sputum TCC >25 million cells/g.
* Clinically significant hepatic impairment or current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Positive HIV, Hepatitis B surface antigen or Hepatitis C antibody within 3 months of screening.
* The subject regularly drinks more than 28 units of alcohol in a week, if male or 21 units per week, if female. One unit of alcohol is defined as a medium (125ml) glass of wine, half a pint (250ml) of beer, or one measure (25ml) of spirits.
* Pregnant and lactating women.
* Asthma considered unstable within 2 months prioir to screening.
* Respiratory Infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within the 4 weeks before screening and led to a change in asthma management, or in the opinion of the Investigator is expected to affect the subjects asthma status or the subjects ability to participate in the study.
* Baseline post-bronchodilator FEV1 <50% predicted (spirometry to be done at screening visit).
* Regular oral prednisone use.
* Subjects who have received therapy with monoclonal antibodies within the proceeding 3 months prior to screening visit.
* Co-morbidities that, in the investigator's opinion may interfere with study including systemic inflammatory conditions such as rheumatoid arthritis.
* Donation of blood in excess of 500 mL within a 56-day period prior to dosing
* Participation in a trial with any drug within 30 days or 5 half-lives (whichever is longer), or participation in a trial with a new chemical entity within 2 months prior to first dose of current study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened but not limited to amphetamines, barbiturates, cocaine, opiates, and cannabinoids.

Subjects who use benzodiazepines or other anxiolytic on a regular basis can be included at the discretion of the investigator and in consultation with the GSK medical monitor.

* Cytochrome P450 3A4 inhibitors including but not limited to antiretrovirals (protease inhibitors) (e.g.indinavir, nelfinavir, ritonavir, saquinavir); imidazole and triazole anti-fungals (e.g.

ketaconazole, itraconazole); macrolide antibiotics (e.g. clarithromycin, erytrhomycin and; telithromycin); calcium channel blockers (diltiazem and verapamil) and nefazodone, 6 weeks before.

* Consumption of seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09-08 (Actual); Primary Completion 2011-08-29 (Actual); Study Completion 2011-08-29 (Actual)

PRIMARY OUTCOMES:
Number of eosinophils (absolute cell count) in induced sputum | Day 10
  Sputum was collected according to the Hargreave/Nair Sputum Induction procedures.Each site performed their sputum analysis locally. Sputum induction for eosinophils was carried out at screening and Day 10. The absolute cell count of eosinophils in induced sputum has been presented.
Number of eosinophils (absolute cell count) in induced sputum following predisone | Day 22
  Sputum was collected according to the Hargreave/Nair Sputum Induction procedures. Each site performed their sputum analysis locally. At Visit 5 (Day 17), all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Sputum induction for eosinophils was carried out at screening and Post Oral Prednisone Visit (Day 22). The absolute cell count of eosinophils in induced sputum has been presented.
Number of eosinophils (percentage count) in induced sputum | Day 10
  Sputum was collected according to the Hargreave/Nair Sputum Induction procedures. Each site performed their sputum analysis locally. Sputum induction for eosinophils was carried out at screening and Day 10. Percentage count of eosinophils in induced sputum has been presented.
Number of eosinophils (percentage count) in induced sputum following prednisone | Day 22
  Sputum was collected according to the Hargreave/Nair Sputum Induction procedures. Each site performed their sputum analysis locally. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Sputum induction for eosinophils was carried out at screening and Post Oral Prednisone Visit (Day 22). Percentage count of eosinophils in induced sputum has been presented.

SECONDARY OUTCOMES:
Number of eosinophils (absolute cell count) in blood | Day 10
  Blood samples for analysis of eosinophils were collected on randomization (Day 1) and end of treatment (Day 10). The absolute cell count for number of eosinophils in blood has been presented.
Number of eosinophils (absolute cell count) in blood following prednisone | Day 22
  At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Blood samples for analysis of eosinophils were collected on randomization (Day 1) and Post Oral Prednisone Visit (Day 22). The absolute cell count for number of eosinophils in blood has been presented.
Eosinophil progenitors in sputum and blood | Day 1, Day 10
  Since only one site collected eosinophil progenitor samples, the data was limited. Sputum and blood eosinophil progenitors analysis (CD34+ and IL5Rα+) was carried out on randomization (Day 1) and end of treatment (Day 10) and Post Oral Prednisone Visit (Day 22).
Chemotactic effect of sputum supernatant on eosinophils | Day 10
  Sputum was collected according to the Hargreave/Nair Sputum Induction procedures. Each site performed their sputum analysis locally. Chemotactic analysis was performed as spontaneous chemotactic activity (Chemotactic activity of the sputum at several dilutions) and Eotaxin-induced chemotaxis (determination in the presence and absence of a single, pre-defined eotaxin concentration spiked into the sputum). In each case the data was a fluorescence intensity which was proportional to the number of migrated cells. The plate-corrected fluorescence intensities were derived by subtracting the mean basal values for each plate from the non-basal individual values on that plate and has been presented as dilution types: neat; 1:03;1:09: 1:27; spiked.
Provocative concentration of methacholine resulting in a 20 percent reduction (PC 20) in forced expiratory volume in 1 second (FEV1). | Day 10
  FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants inhaled doubling increments of methacholine until a >=20 percent fall in FEV1 from the saline value was achieved.
Change from baseline in forced expiratory volume in 1 second (FEV1) | From Baseline (Day 1) to Day 10 and Day 17
  FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Spirometry using FEV1 was performed at Day 1 (visit 2), Day 10 (visit 4), Day 17 (visit 5). Baseline was defined as value at Day 1 (visit 2). Change from baseline was calculated by subtracting the baseline value from the post-randomization values at Days 10 and 17.
Change from baseline in FEV1 following prednisone | Baseline (Day 1) to Day 22
  FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Spirometry using FEV1 was performed at Day 22 (visit 6). Baseline was defined as value at Day 1 (visit 2). Change from baseline was calculated by subtracting the baseline value from the post-randomization value at Days 22.
Assessment of asthma stability using Asthma Control Questionnaire (ACQ) | Day 1 and Day 10
  The ACQ consists of seven questions that were scored on a seven-point scale from 0 to 6. The response options for all these questions consisted of a 0 (no impairment/limitation) to 6 (total impairment/ limitation) scale. The ACQ score was derived as the mean of the seven questions, where the mean score ranged from 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicated severity. ACQ was set to missing if any of the seven questions had a missing response. Assessments were carried out on Day 1 (visit 2) and Day 10 (visit 4).
Assessment of vital sign systolic blood pressure (SBP) and diastolic blood pressure (DBP) | Upto Day 22
  Vital signs measurements included SBP and DBP assessments carried out on Day 1 (visit 2), Day 7 (visit 3), Day 10 (visit 4), Day 17 (visit 5) & Day 22 (visit 6).
Assessment of vital sign heart rate | Upto Day 22
  Vital signs measurements included heart rate assessments carried out on Day 1 (visit 2), Day 7 (visit 3), Day 10 (visit 4), Day 17 (visit 5) & Day 22 (visit 6).
Number of participants with abnormal electrocardiogram (ECG) findings | Day 1 and Day 10
  Twelve-lead ECGs were recorded in the supine position at the screening, randomization (Day 1) and end of treatment (Day 10) prior to administration of the dose. An automatic ECG machine was used to calculate the heart rate and measure PR, QRS, QT, and QTc intervals. The abnormal findings were categorized as abnormal- not clinically significant (A-NCS) and Abnormal - clinically significant (A-CS).
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From start of first dose of study drug, Day 1 to upto Day 17
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new/exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury. Assessments were carried out at Day 1 (visit 2), Day 7 (visit 3), Day 10 (visit 4), Day 17 (visit 5).
Number of participants with AEs and SAEs following prednisone | From start of first dose of study drug Day 1 up to follow-up Day 22
  An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom/disease (new/exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant/require medical/surgical intervention. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Spirometry using FEV1 was performed at Day 22 (visit 6).
Assessment of clinical chemistry parameters albumin and Total protein | Day 10
  Blood samples for clinical laboratory evaluation (chemistry parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The chemistry parameters included assessments for albumin, and total protein. Assessments were performed at screening and Day 10 (visit 4).
Assessment of clinical chemistry parameters albumin and Total protein following prednisone | Day 22
  Blood samples for clinical laboratory evaluation (chemistry parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The chemistry parameters included assessments for albumin, and total protein. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessments were performed at screening and Day 22 (visit 6).
Assessment of clinical chemistry parameters creatinine and uric acid | Day 10
  Blood samples for clinical laboratory evaluation (chemistry parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The chemistry parameters included assessments for creatinine and uric acid. Assessments were performed at screening and Day 10.
Assessment of clinical chemistry parameters creatinine and uric acid following prednisone | Day 22
  Blood samples for clinical laboratory evaluation (chemistry parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The chemistry parameters included assessments for creatinine and uric acid. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessments were performed at screening and Day 22 (visit 6).
Assessment of hematology parameters basophils, eosinophils, lymphocytes, monocytes, total absolute neutrophil count (TANC),platelet count (PC),white blood cell count (WBC) | Day 10
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessments for basophils, eosinophils, lymphocytes, monocytes, TANC, PC and WBC. Assessments were performed at screening and Day 10 (visit 4).
Assessment of hematology parameters basophils, eosinophils, lymphocytes, monocytes, TANC, PC, WBC following prednisone | Day 22
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessments for basophils, eosinophils, lymphocytes, monocytes, TANC, PC and WBC. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessments were performed at screening and Day 22 (visit 6).
Assessment of clinical chemistry parameters calcium, chloride ,carbon dioxide content/bicarbonate, glucose, potassium, sodium ,Urea /Blood urea nitrogen (BUN) | Day 10
  Blood samples for clinical laboratory evaluation (chemistry parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The chemistry parameters included assessments for calcium, chloride ,carbon dioxide content/bicarbonate, glucose, potassium, sodium ,Urea /BUN. Assessments were performed at screening and Day 10 (visit 4).
Assessment of clinical chemistry parameters calcium, chloride ,carbon dioxide content/bicarbonate, glucose, potassium, sodium ,Urea / BUN following prednisone | Day 22
  Blood samples for clinical laboratory evaluation (chemistry parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The chemistry parameters included assessments for calcium, chloride ,carbon dioxide content/bicarbonate, glucose, potassium, sodium ,Urea /BUN. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessments were performed at screening and Day 22 (visit 6).
Assessment of hematology parameters hemoglobin and mean corpuscle hemoglobin concentration (MCHC) | Day 10
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessments for hemoglobin and MCHC. Assessments were performed at screening and Day 10 (visit 4).
Assessment of hematology parameters hemoglobin and MCHC following prednisone | Day 22
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessments for hemoglobin and MCHC. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessments were performed at screening and Day 22 (visit 6).
Assessment of hematology parameter hematocrit | Day 10
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessment for hematocrit. Assessments were performed at screening and Day 10 (visit 4).
Assessment of hematology parameter hematocrit following prednisone | Day 22
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessment for hematocrit. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessments were performed at screening and Day 22 (visit 6).
Assessment of hematology parameter mean corpuscle hemoglobin (MCH) | Day 10
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessment for MCH. Assessments were performed at screening and Day 10 (visit 4).
Assessment of hematology parameter MCH following prednisone | Day 22
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessment for MCH. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessments were performed at screening and Day 22 (visit 6).
Assessment of hematology parameter mean corpuscle volume (MCV) | Day 10
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessment for MCV. Assessments were performed at screening and Day 10 (visit 4).
Assessment of hematology parameter MCV following prednisone | Day 22
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessment for MCV. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessments were performed at screening and Day 22 (visit 6).
Assessment of hematology parameter red blood cell count (RBC) | Day 10
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessment for RBC. Assessments were performed at screening and Day 10 (visit 4).
Assessment of hematology parameter RBC following prednisone | Day 22
  Blood samples for clinical laboratory evaluation (hematology parameters) were obtained at screening and follow-up only. Samples were collected following an overnight fast when feasible. The hematology parameter included assessment for RBC. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessments were performed at screening and Day 22 (visit 6).
Assessment of liver function tests (LFTs) alkaline phosphatase, alanine amino transferase (ALT), aspartate amino transferase (AST) and gamma glutamyl transferase (GGT) as a measure of monitoring liver toxicity | Upto Day 17
  LFTS included alkaline phosphatase, ALT, AST and GGT as a measure of monitoring liver toxicity. Assessment were carried out at Screening, Day 1 (visit 2), Day 7 (visit 3), Day 10 (visit 4), Day 17 (visit 5).
Assessment of LFTs alkaline phosphatase, ALT, AST and GGT as a measure of monitoring liver toxicity following prednisone | Day 22
  LFTS included alkaline phosphatase, ALT, AST and GGT as a measure of monitoring liver toxicity. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessment were carried out at Screening and Day 22 (visit 6).
Assessment of LFTs direct bilirubin and total bilirubin as a measure of monitoring liver toxicity. | Upto Day 17
  LTFS included direct bilirubin and total bilirubin as a measure of monitoring liver toxicity. Assessment were carried out at Screening, Day 1 (visit 2), Day 7 (visit 3), Day 10 (visit 4), Day 17 (visit 5).
Assessment of LFTs direct bilirubin and total bilirubin as a measure of monitoring liver toxicity following prednisone | Day 22
  LTFS included direct bilirubin and total bilirubin as a measure of monitoring liver toxicity. At Visit 5, all participants were given 30 mg oral daily prednisone for 5 days and participants returned to clinic at a Post Oral Prednisone Visit (Visit 6) at Day 22. Assessment were carried out at Screening and Day 22 (visit 6).
Assessment of plasma concentrations of GW766994 Pre-dose Day 7 (Visit 3) and Day 10 (Visit 4) | Pre-dose Day 7 (Visit 3) and Day 10 (Visit 4)
  Pharmacokinetic samples were collected from each participant according to the sample schedule on Day 2 (visit 3) and 7 (visit 4). Concentrations of GW766994 in plasma have been and summarized by treatment group and nominal time ( i.e. pre-dose).
Assessment of plasma concentrations of GW766994 1 hours post-dose on Day 1 (Visit 2), Day 7 (Visit 3) and Day 10 (Visit 4) | Day 1 (Visit 2), Day 7 (Visit 3) and Day 10 (Visit 4)
  Pharmacokinetic samples were collected from each participant according to the sample schedule on Day 1 (visit 2), Day 2 (visit 3) and Day 7 (visit 4). Concentrations of GW766994 in plasma have been and summarized by treatment group and nominal time ( i.e. 1 hour post- dose).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register